CLINICAL TRIAL: NCT05237271
Title: Establishing Clinical Utility Evidence to Support Coverage and Reimbursement for SomaLogic's Cardiovascular Disease in Type 2 Diabetes Test: A CPV® Randomized Controlled Trial
Brief Title: Clinical Utility Trial for the SomaLogic CVD-T2D Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: SomaLogic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00058735
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Control group treats their simulated patients using standard practice and have no introduction to the new SomaLogic test.
- Intervention Group 1 (Experimental): Intervention group 1 will receive educational materials on the single cardiovascular disease in type 2 diabetes risk score. They will then be forced to used the risk score for their simulated patients, which will allow us to assess how the risk score may improve clinical practice and reduce variation.
  Interventions: Other: Educational Materials on the Cardiovascular Disease in Type 2 Diabetes (CVD-T2D)
- Intervention Group 2 (Experimental): Intervention group 2 will receive educational materials on the cardiovascular disease in type 2 diabetes (CVD-T2D) risk score as well as the panel of metabolic scores. They will then be forced to used the CVD-T2D score and the metabolic panel scores for their simulated patients, which will allow us to assess how the risk score may improve clinical practice and reduce variation.
  Interventions: Other: Educational Materials on the Cardiovascular Disease in Type 2 Diabetes (CVD-T2D); Other: Educational Materials on the CVD-T2D and Bundled Metabolic Panel

INTERVENTIONS:
Other: Educational Materials on the Cardiovascular Disease in Type 2 Diabetes (CVD-T2D) — Educational Materials will detail the diagnostic tests in question. This CVD-T2D will provide a numerical risk score for the likelihood of patients with type 2 diabetes to have a cardiovascular event in the next 4 years.
  Arms: Intervention Group 1; Intervention Group 2
Other: Educational Materials on the CVD-T2D and Bundled Metabolic Panel — Educational Materials will detail the diagnostic tests in question.his CVD-T2D will provide a numerical risk score for the likelihood of patients with type 2 diabetes to have a cardiovascular event in the next 4 years. The bundled metabolic scores will provide insight into the patient's current metabolic conditions.
  Arms: Intervention Group 2

SUMMARY:
QURE will use its CPV technology in a randomized controlled trial to measure how SomaLogic's diagnostic test (the Cardiovascular Disease in Type 2 Diabetes) changes clinical practice and improves patient outcomes.

DETAILED DESCRIPTION:
SomaLogic has developed a pioneering technology, the SomaScan® Platform, the first and only platform, that simultaneously measures 7,000 proteins. The company's technology is based on proprietary aptamers, called SOMAmers®, which can measure these unique proteins with high sensitivity and specificity across a large dynamic range. Using over 60,000 samples, artificial intelligence and machine learning powered bioinformatics algorithms have created 12 SomaSignal™ tests. The Cardiovascular Disease in Type 2 Diabetes (CVD-T2D) Test result produces risk score for developing cardiovascular events such as heart attacks, strokes, heart failure, or cardiovascular death within 4 years, with median time to event of 1.7 years across the different risk categories. SomaSignal™ testing has the potential to effectively risk-stratify patients, determine disease prognosis, and elucidate disease drivers for clinicians. Analytic and clinical validity findings, using this patented technology, have already been published by the company or collaborators in scientific and clinical manuscripts.

SomaLogic is looking to understand if the test, when used by practitioners, helps clinicians determine cardiovascular risk status and achieve better care for patients with diabetes. To achieve this goal, SomaLogic is looking for an established, innovative approach to gather high-quality prospective clinical utility data in as short a time as possible. Determining the clinical utility of the SomaSignal tests will be essential to increase access to the test and is required to gain coverage and reimbursement.

Accordingly, this study will collect high-quality randomized controlled data from a nationally representative sample of practicing primary care physicians and cardiologists. To first determine how these physicians currently manage cardiovascular risk factors in patients with Type 2 Diabetes (T2DM) and then to determine if introducing the test results of the CVD-T2D test will change their clinical decision making. Data from this study will better illuminate which use case is best served by SomaSignal testing (and thus the greatest clinical utility) and what physician characteristics (e.g., age, practice setting, training) are associated with these practice changes.

This study uses simulated patient cases, called Clinical Performance and Value vignettes (CPVs), a proven methodology that is widely used to rapidly measure physician care decisions. CPVs are a unique and scalable tool that standardizes practice measurement by having all providers care for the same (virtual) patients. With all providers caring for the same patients, the CPVs generate unbiased data that yields powerful insights into clinical decision making and how these decisions change with the introduction of a new product or solution. Data from the CPVs demonstrates the presence or absence of the clinical utility of a diagnostic test. The results, positive or negative, are published in peer-reviewed literature and if they are positive, favorably impact coverage and reimbursement decisions.

The primary goal will be to determine whether informing clinicians of the CVD-T2D test results leads to changes in prescriptions and/or medical management of virtual participants with T2D in concordance with CVD in Type 2 Diabetes results compared with virtual participants whose physicians are not informed of the test results.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified primary care physicians or cardiologist for at least two years
2. Averaging at least 20 hours per week of clinical and patient care duties over the last six months
3. Routinely evaluate patients with diabetes mellitus in their practice
4. Practicing in the U.S.
5. English speaking
6. Access to the internet
7. Informed, signed and voluntarily consented to be in the study

Exclusion Criteria:

1. Non-English speaking
2. Practicing in an academic setting
3. Unable to access the internet
4. Not practicing in the U.S.
5. Not averaging at least 20 hours per week of clinical or patient care duties over the last six months
6. Previous exposure to the CVD-T2D test
7. Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
CPV-measured clinical score difference | 12 Months
  Difference-in-differences regression analysis between the control and the intervention groups' physicial exam, workup, diagnosis, and treatment cardiovascular risk in patients with type 2 diabetes, as measured by the participants diagnostic and treatment CPV case domain scores. In each CPV, participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum from 0 to a high potential score of up to 100 percent in each domain, where higher scores mean better outcomes. We will measure the overall change in the evidence-based physician behavior including referrals, utilization of cardioprotective medications, right heart catherization and echocardiography, in the CPV patient simulations.
CPV-measured cost difference | 12 Months
  Change in cost of related care for cardiovascular risks in patients with diabetes mellitus when comparing the control to the intervention group. (This cost is modeled in part by measuring differential rates of medical interventions selected by each arm and multiplying by average Medicare reimbursement rates for these interventions. The cost is also modeled by examining average per annum costs for patients suffering from diabetes mellitus and multiplying by the percent of patients whose workup and interventions for cardiovascular risks are significantly reduced following the intervention.)

SECONDARY OUTCOMES:
CPV-measured baseline clinical variation levels | 12 Months
  Participants completing the simulated cases, or CPVs, receive scores based upon the quality of care they provide. This measure will assess the baseline levels of variation in the care of pain patients among all participants, including by use case types. We will measure the baseline levels of variation in the assessment, recognition, and management of cardiovascular risks in patients with diabetes mellitus among all participants.
CPV-measured Assessment of use case types | 12 Months
  Difference in the overall, and the diagnostic and treatment quality scores between control and intervention participants. Diagnostic and treatment scores are calculated as the percent correct on CPVs, and the overall score is a average score of the subcategory scores (percent correct). This will be examined for each of the use cases to determine in which case(s) CPV scores most improved.

CONTACTS AND LOCATIONS:
Overall Officials: John W Peabody, MD, PhD, Principal Investigator — QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

REFERENCES:
- [Derived] Peabody JW, Paculdo D, de Belen E, Ganesan D, Cooney I, Trujillo N. Clinical utility of a novel test for assessing cardiovascular disease risk in type 2 diabetes: a randomized controlled trial. Diabetol Metab Syndr. 2023 Jul 13;15(1):155. doi: 10.1186/s13098-023-01122-w. PMID 37438853